CLINICAL TRIAL: NCT03368924
Title: Implication of the Oxydative Stress in the Pathophysiology of Sickle Cell Anemia: Vaso-occlusive Crises, Anti Bande 3 Antibodies Levels, Red Blood Cell Oxidation
Brief Title: Implication of the Oxydative Stress in the Pathophysiology of Sickle Cell Anemia:
Acronym: STRESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de la Guadeloupe (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RBM-PAP-2012/47
Record Dates: First submitted 2017-12-01; First posted 2017-12-11 (Actual); Last update posted 2017-12-11 (Actual); Status verified 2017-11

CONDITIONS: Sickle Cell Disease
Keywords: sickle cell anemia red blood cell oxidation; vaso-occlusive crises; anti bande 3 antibodies; red blood cell oxidation
MeSH Terms: conditions — Anemia, Sickle Cell; Vaso-Occlusive Crises

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SCA patients (SS genotype) (Other): * To compare the level of anti band 3 antibodies in steady state and during vaso-occlusive crises in SCA patients.
  * To assess the relationship between level of biomarkers of oxidation of SS RBCs, altered hemorheological parameters, biomarkers of cellular activation (microparticles) and anti band 3 antibodies rate, taking into account the alpha-globin genes status.
  * To study the relationship between level of anti band 3 antibodies and severity of these VOC using an index of clinical severity (IS2) calculated at the end of SCA patients hospitalization for VOC.
  * To study early clinical (including the activity of the autonomic nervous system activity) and biological items to evaluate the relationship between these items and severity of VOC.
  Interventions: Other: SCA patients (SS genotype)

INTERVENTIONS:
Other: SCA patients (SS genotype) — The clinical data relative to the patients will be collected in each of these stages (CVO, basic state).
  Besides, to estimate the severity of the CVO, we shall use an index of severity of the episode ( IS2) adapted from the one who was validated by our group to stratify the severity of vasoocclusifs episodes at the drepanocytic child SS.
  Main clinical parameters: taken of analgesic at home (level), temperature in the admission, SaO2 in the admission, number of painful sites, thoracic pain with or without associated cough, score EVA in the entrance, feeling of the patient of bigger gravity of the CVO with regard to its crises previous, heart rate to the admission, … Main biological parameters: rate of leukocytes, of polynucléaires neutrophiles, of réticulocytes, Lactate déshydrogénase, of haemoglobin, C-reactive Protein … The biological data can be studied according to their raw rate or according to their difference with their basic value (in the stable state).

SUMMARY:
Despite important advances in the current understanding of sickle cell vaso-occlusion, the basis of its control and prevention remain partially unknown. The primary purpose is to test the hypothesis of a control of the sickle cell vaso-cocclusive (VOC) process by the anti band 3 antibodies by assessing the level of these antibodies in the steady state and during the crises in SCA patients. To assess the relationship between the level of band 3 antibodies, the oxidation status, the expression of microparticles and the hemorheological alterations of the sickle red cells (SS RBs), the severity of VOC.

DETAILED DESCRIPTION:
Although oxidative stress is not the primary aetiology of SCA, oxidative damage could in part account for pathophysiological mechanisms leading to sickle vaso-occlusion, in which anti bande 3 antibodies might play a role. Bande 3 is a protein belonging to red blood cells. These anti bande 3 antibodies are producted when after oxidative damage, a hidden site of bande 3 is revealed. In preliminary data, the Cuban partner of this study showed a significative difference between their level in patients, during steady state and vaso-occlusive crises. Our clinical question is to determine if a decrease of these antibodies, could participate in the occurrence of the crises. Therapeutic strategies aimed to counteract oxidative abnormalities might alleviate this still nowadays unknown mechanisms disease progression.

Band 3 protein which belongs to the anionic interchanger is the main erythrocyte membrane protein, present in about 1.2 x 106 copies per cell. Under certain conditions, band 3 protein modifications in the human erythrocyte membrane surface lead to band 3 aggregates. These modifications are mostly due to oxidative insults that gradually accumulate during red blood cell lifespan. Band 3 clusters on the SS RBCs produce two significant changes: first, these cells acquire an adhesive nature; second, band 3 aggregates are recognized by natural band 3 antibodies. Several studies have shown that band 3 peptides are able to inhibit the adherence of SS RBCs to endothelial cells. This suggests possible participation of band 3 antibodies in the aethiology as well as in the prevention of VOC in SCA. Oxidant damage in RBCs may contribute to the circulatory disorders by affecting their flow properties i.e. their deformability, aggregability and adherence to endothelial cells. Therefore, in parallel of the study of the evaluation of the role of anti bande 3 antibodies in VOC occurrence and severity, the investigators will explore the involvement of oxidative stress on the rheological properties of SSRBCs (deformability and aggregability),

ELIGIBILITY:
Inclusion Criteria:

- adults ≥ 18 years old SCA patients (SS genotype) hospitalized for bone VOC with single or multifocal localizations.

Exclusion Criteria:

* chronic transfusion therapy or recent blood transfusion (less than 3 months before the current VOC or the state defined "steady-state" in SCA);
* severe chronic renal failure; liver failure;
* autoimmune disease;
* viral hepatitis; HIV seropositivity;
* pregnancy or breast feeding;
* patients already engaged in another therapeutic clinical research protocol; - non-compliant patients to usual care;
* patients unable to give their consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2013-04-09 (Actual); Primary Completion 2015-09-19 (Actual); Study Completion 2015-09-19 (Actual)

PRIMARY OUTCOMES:
To compare the level of anti band 3 antibodies in steady state and during vaso-occlusive crises in SCA patients. | Through study completion, an average of 3 years
  Dosage of anti band 3 antibody during the steady state and the VOC

SECONDARY OUTCOMES:
To assess the relationship between level of biomarkers of oxidation of SS RBCs, altered hemorheological parameters, biomarkers of cellular activation (microparticles) and anti band 3 antibodies rate, taking into account the alpha-globin genes status | Through study completion, an average of 3 years
  Dosage of Parameters hémorhéologiques Dosage of the circulating microparticles Assessment of the level of oxidation of red blood cells
To study the relationship between level of anti band 3 antibodies and severity of these VOC using an index of clinical severity (IS2) calculated at the end of SCA patients hospitalization for VOC. | Through study completion, an average of 3 years
  Dosage of anti band 3 antibody during the VOC Index of clinical severity (IS2)
To study early clinical (including the activity of the autonomic nervous system activity) and biological items to evaluate the relationship between these items and severity of VOC. | Through study completion, an average of 3 years
  Dosage of Parameters hémorhéologiques Dosage of the circulating microparticles Assessment of the level of oxidation of red blood cells clinical evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie LEMONNE, Doctor specializing in SCA, Principal Investigator — Hospital University Center of Pointe-à-Pitre
Locations (1):
- Hospital University Center of Pointe-à-Pitre, Pointe-à-Pitre, Guadeloupe